CLINICAL TRIAL: NCT00129181
Title: A Single-blinded Assessment of the Short-term Effects of Cabergoline vs. Carbidopa/Levodopa on SPECT Dopamine Transporter Density in Out-patient Subjects With Parkinson's Disease
Brief Title: Study of the Effects of Dopaminergic Medications on Dopamine Transporter Density in Subjects With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Pfizer (Industry); GE Healthcare (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AMAD001
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Parkinson Disease; Parkinsonian Syndrome
Keywords: parkinson; brain imaging; diagnosis
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Disease | interventions — Cabergoline; carbidopa, levodopa drug combination; ioflupane

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cabergoline — Approximately 120 Parkinson's disease subjects will be randomized to receive either carbidopa/levodopa, cabergoline or no treatment during a twelve week period. Subjects will undergo SPECT imaging with DATscan at screening and after 12 weeks. After twelve weeks carbidopa/levodopa and cabergoline treatment will be withdrawn and all subjects will undergo SPECT imaging with DATscan after 8 weeks (20 weeks after baseline).
Drug: carbidopa/levodopa — Approximately 120 Parkinson's disease subjects will be randomized to receive either carbidopa/levodopa, cabergoline or no treatment during a twelve week period. Subjects will undergo SPECT imaging with DATscan at screening and after 12 weeks. After twelve weeks carbidopa/levodopa and cabergoline treatment will be withdrawn and all subjects will undergo SPECT imaging with DATscan after 8 weeks (20 weeks after baseline).
Procedure: DATscan and SPECT imaging — Approximately 120 Parkinson's disease subjects will be randomized to receive either carbidopa/levodopa, cabergoline or no treatment during a twelve week period. Subjects will undergo SPECT imaging with DATscan at screening and after 12 weeks. After twelve weeks carbidopa/levodopa and cabergoline treatment will be withdrawn and all subjects will undergo SPECT imaging with DATscan after 8 weeks (20 weeks after baseline).

SUMMARY:
This study investigates whether there is a change in 123iodine-2ß- carbomethoxy-3ß-(4-iodophenyl) tropane ([123I]ß-CIT) uptake after short-term treatment with levodopa compared to either dopamine agonist or placebo.

DETAILED DESCRIPTION:
This is a multi-center, open-label study of short-term treatment with levodopa or cabergoline on striatal DATscan uptake in early Parkinson's disease. Approximately 120 Parkinson's disease subjects will be randomized to receive either carbidopa/levodopa, cabergoline or no treatment during a twelve week period. Subjects will undergo SPECT imaging with DATscan at screening and after 12 weeks. After twelve weeks carbidopa/levodopa and cabergoline treatment will be withdrawn and all subjects will undergo SPECT imaging with DATscan after 8 weeks (20 weeks after baseline).

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged 40 years or older.
* Written informed consent is obtained.
* Subjects have a clinical diagnosis of idiopathic Parkinson's disease.
* Hoehn and Yahr stages for subjects are I-II.

Exclusion Criteria:

* The subject has atypical or drug-induced Parkinson's disease.
* The subject has dementia.
* The subject has clinically significant abnormal laboratory values, and/or clinically significant or unstable medical or psychiatric illness.
* The subject is pregnant.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To determine the influence of short-term levodopa therapy on dopamine transporter density in early Parkinson's disease | 1 year

SECONDARY OUTCOMES:
To determine the influence of short-term treatment with cabergoline on dopamine transporter density in early Parkinson's disease | 1 year
To further develop the AMADEUS consortium, a collaboration of clinical-imaging SPECT DAT sites able to obtain data using comparable techniques and transmit imaging to a central analysis site | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Marek, MD, Principal Investigator — The Institute for Neurodegenerative Disorders; John P Seibyl, MD, Principal Investigator — The Institute for Neurodegenerative Disorders
Locations (9):
- Austria (2):
  - Department of Neurology, Innsbruck Medical University, Innsbruck
  - Neurological Department, Wilhelminenspital, Vienna
- Germany (3):
  - Dept. of Neurology, University of Leipzig, Leipzig
  - Dept. of Neurology Marburg, Phillips-Univ., Marburg
  - Ambulanz für Bewegungsstörungen, Neurologische Poliklinik, München
- Italy (3):
  - University of Catania-Department of Neurosciences, Catania
  - Parkinson Institute Milan, Milan
  - Department of Neurological Sciences-University of Napoli, Naples
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

REFERENCES:
- [Background] Ahlskog JE. Slowing Parkinson's disease progression: recent dopamine agonist trials. Neurology. 2003 Feb 11;60(3):381-9. doi: 10.1212/01.wnl.0000044047.58984.2f. PMID 12580184
- [Background] Ahlskog JE, Uitti RJ, O'Connor MK, Maraganore DM, Matsumoto JY, Stark KF, Turk MF, Burnett OL. The effect of dopamine agonist therapy on dopamine transporter imaging in Parkinson's disease. Mov Disord. 1999 Nov;14(6):940-6. doi: 10.1002/1531-8257(199911)14:63.0.co;2-y. PMID 10584667
- [Background] Brucke T, Asenbaum S, Pirker W, Djamshidian S, Wenger S, Wober C, Muller C, Podreka I. Measurement of the dopaminergic degeneration in Parkinson's disease with [123I] beta-CIT and SPECT. Correlation with clinical findings and comparison with multiple system atrophy and progressive supranuclear palsy. J Neural Transm Suppl. 1997;50:9-24. PMID 9120429
- [Background] Fahn S. Is levodopa toxic? Neurology. 1996 Dec;47(6 Suppl 3):S184-95. doi: 10.1212/wnl.47.6_suppl_3.184s. No abstract available. PMID 8959987
- [Background] Guttman M, Stewart D, Hussey D, Wilson A, Houle S, Kish S. Influence of L-dopa and pramipexole on striatal dopamine transporter in early PD. Neurology. 2001 Jun 12;56(11):1559-64. doi: 10.1212/wnl.56.11.1559. PMID 11402115
- [Background] Innis RB, Seibyl JP, Scanley BE, Laruelle M, Abi-Dargham A, Wallace E, Baldwin RM, Zea-Ponce Y, Zoghbi S, Wang S, et al. Single photon emission computed tomographic imaging demonstrates loss of striatal dopamine transporters in Parkinson disease. Proc Natl Acad Sci U S A. 1993 Dec 15;90(24):11965-9. doi: 10.1073/pnas.90.24.11965. PMID 8265656
- [Background] Innis RB, Marek KL, Sheff K, Zoghbi S, Castronuovo J, Feigin A, Seibyl JP. Effect of treatment with L-dopa/carbidopa or L-selegiline on striatal dopamine transporter SPECT imaging with [123I]beta-CIT. Mov Disord. 1999 May;14(3):436-42. doi: 10.1002/1531-8257(199905)14:33.0.co;2-j. PMID 10348466
- [Background] Little KY, Gorebig J, Carroll FI, Mapili J, Meador-Woodruff JH. Lack of dopamine receptor agonists effect on striatal dopamine transporter binding sites. Brain Res. 1996 Dec 2;742(1-2):313-6. doi: 10.1016/s0006-8993(96)01033-5. PMID 9117410
- [Background] Marek K, Innis R, van Dyck C, Fussell B, Early M, Eberly S, Oakes D, Seibyl J. [123I]beta-CIT SPECT imaging assessment of the rate of Parkinson's disease progression. Neurology. 2001 Dec 11;57(11):2089-94. doi: 10.1212/wnl.57.11.2089. PMID 11739831
- [Background] Morrish PK, Rakshi JS, Bailey DL, Sawle GV, Brooks DJ. Measuring the rate of progression and estimating the preclinical period of Parkinson's disease with [18F]dopa PET. J Neurol Neurosurg Psychiatry. 1998 Mar;64(3):314-9. doi: 10.1136/jnnp.64.3.314. PMID 9527140
- [Background] Nurmi E, Bergman J, Eskola O, Solin O, Hinkka SM, Sonninen P, Rinne JO. Reproducibility and effect of levodopa on dopamine transporter function measurements: a [18F]CFT PET study. J Cereb Blood Flow Metab. 2000 Nov;20(11):1604-9. doi: 10.1097/00004647-200011000-00010. PMID 11083235
- [Background] Parkinson Study Group. Dopamine transporter brain imaging to assess the effects of pramipexole vs levodopa on Parkinson disease progression. JAMA. 2002 Apr 3;287(13):1653-61. doi: 10.1001/jama.287.13.1653. PMID 11926889
- [Background] Fahn S; Parkinson Study Group. Does levodopa slow or hasten the rate of progression of Parkinson's disease? J Neurol. 2005 Oct;252 Suppl 4:IV37-IV42. doi: 10.1007/s00415-005-4008-5. PMID 16222436
- [Background] Rioux L, Frohna PA, Joyce JN, Schneider JS. The effects of chronic levodopa treatment on pre- and postsynaptic markers of dopaminergic function in striatum of parkinsonian monkeys. Mov Disord. 1997 Mar;12(2):148-58. doi: 10.1002/mds.870120204. PMID 9087972
- [Background] Schapira AH. Dopamine agonists and neuroprotection in Parkinson's disease. Eur J Neurol. 2002 Nov;9 Suppl 3:7-14. doi: 10.1046/j.1468-1331.9.s3.9.x. PMID 12464116
- [Background] Whone AL, Watts RL, Stoessl AJ, Davis M, Reske S, Nahmias C, Lang AE, Rascol O, Ribeiro MJ, Remy P, Poewe WH, Hauser RA, Brooks DJ; REAL-PET Study Group. Slower progression of Parkinson's disease with ropinirole versus levodopa: The REAL-PET study. Ann Neurol. 2003 Jul;54(1):93-101. doi: 10.1002/ana.10609. PMID 12838524
- [Background] Wooten GF. Agonists vs levodopa in PD: the thrilla of whitha. Neurology. 2003 Feb 11;60(3):360-2. doi: 10.1212/wnl.60.3.360. No abstract available. PMID 12578913